CLINICAL TRIAL: NCT01208220
Title: The Effects of Collagenase Santyl Ointment and Negative Pressure Wound Therapy(Npwt) for the Treatment of Chronic Pressure Ulcers.
Brief Title: Effectiveness Study of Santyl Ointment to Treat Pressure Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment of qualified subjects
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Healthpoint (Industry)
Responsible Party: Principal Investigator, Dr. Stanley McCallon, Assistant Professor - School of Physical Therapy, Louisiana State University Health Sciences Center Shreveport
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Healthpoint-123-Collagenase
Record Dates: First submitted 2010-04-16; First posted 2010-09-23 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Pressure Ulcer; Soft Tissue Necrosis Lower Limb
Keywords: Collagenase Santyl; Enzymatic debridement; maintenance debridement; VAC; NPWT
MeSH Terms: conditions — Pressure Ulcer | interventions — Negative-Pressure Wound Therapy; Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Negative pressure wound therapy (Active Comparator): NPWT changed TIW
  Interventions: Device: Negative Pressure Wound Therapy
- NPWT plus Collagenase Ointment (Experimental): Collagenase applied TIW with NPWT
  Interventions: Biological: Collagenase Ointment

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — NPWT changed 3 times weekly
  Other Names: NPWT
  Arms: Negative pressure wound therapy
Biological: Collagenase Ointment — Apply TIW
  Arms: NPWT plus Collagenase Ointment

SUMMARY:
Researchers at LSUHSC-S hope to learn the effects of the combination of a medication and a device which by themselves are effective for the treatment of wounds.

You are being asked to take part in this study because you have a wound on your body which has not responded to standard treatments.

The researchers will be studying whether the combination of two treatments will make wounds heal faster. For those in study, the investigators will treat them with a vacuum device on their wound. Also, some of the people in the study will receive a special ointment and researchers will use special tests to determine if the two treatments together are working better than just one treatment alone.

DETAILED DESCRIPTION:
Evaluate the effectiveness of Collagenase Santyl ointment when used in conjunction with NPWT for the treatment of chronic pressure ulcers and determine whether the addition of Collagenase Santyl ointment has a positive effect on wound healing. Through volumetric changes and histological evaluation, we wish to test the hypothesis that the application of Collagenase Santyl ointment in conjunction with NPWT facilitates improved wound healing and mitigates some potentially harmful effects of NPWT alone (e.g. pain with dressing removal and tissue ingrowth

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 year-old competent adults in inpatient setting (no prisoners, mentally ill, or children)
* Pressure ulcers to pelvis/abdomen/trunk and or upper extremities which have been refractory to prior treatment interventions and contain less than or equal to 25% necrotic tissue in wound bed (as percentage of total surface area)

Exclusion Criteria:

* Lower extremity/foot wounds related to arterial insufficiency, incarcerated individuals, patients with untreated osteomyelitis, uncorrected coagulopathy, malignancy, sensitivity to collagenase, wounds with evidence of clinical infection (via swab culture or punch biopsy)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley K McCallon, DPT, Principal Investigator — LSUHSC professor
Locations (1):
- LSU Health Sciences Center, Shreveport, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Large acute care hospital
Groups:
- Negative Pressure Wound Therapy: NPWT alone for treatment of pressure ulcer
  NPWT - VAC : Vacuum Assisted Closure at 125 mm of negative pressure continuous, dressing changed three times weekly
- Santyl Ointment and NPWT: Enzymatic debriding ointment used in conjunction with negative pressure wound therapy
  Collagenase Santyl : Topical enzyme applied to wound tissue
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy | Santyl Ointment and NPWT
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure Wound Therapy | Santyl Ointment and NPWT | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (0) | 57 (0) | 54 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Removal of Harmful Fluids in the Wound Tissue
Time Frame: 2 weeks into study
Measure: Number; unit: percentage of cytotoxins removed
Arm/Group | Negative Pressure Wound Therapy | Santyl Ointment and NPWT
Number analyzed (Participants) | 1 | 1
percentage of cytotoxins removed | 0 | 0

2. Primary Outcome: Quicker Filling of the Wound With Good Tissue (vs. Treatment With NPWT Alone)
Time Frame: 2 weeks into study
Measure: Number; unit: Percentage of red granulation tissue
Arm/Group | Negative Pressure Wound Therapy | Santyl Ointment and NPWT
Number analyzed (Participants) | 1 | 1
Percentage of red granulation tissue | 80 | 75

ADVERSE EVENTS:
Arm/Group | Negative Pressure Wound Therapy | Santyl Ointment and NPWT
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
No adverse events noted or reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No